CLINICAL TRIAL: NCT03081676
Title: The Effect of GIP and GLP-1 on Insulin and Glucagon Secretion in Patients With HNF1A-diabetes Treated With or Without Sulphonylurea
Acronym: HNF1A-Clamp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Alexander Christensen, MD, PhD student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-16038140
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Maturity-Onset Diabetes of the Young, Type 3
Keywords: Maturity-Onset Diabetes of the Young, Type 3; Glucose-dependent insulinotropic peptide; Glucagon-like-peptide 1; Dipeptidyl peptidase 4; Glimepiride; Sulphonylurea; Glucose clamp; Hepatocyte nuclear factor 1 alpha
MeSH Terms: conditions — Maturity-Onset Diabetes of the Young, Type 3 | interventions — glimepiride; Tablets; Glucagon-Like Peptide 1; Incretins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Glimepiride + GIP (Active Comparator): Tablet Glimepiride + infusion of GIP
  Interventions: Drug: Glimepiride 1Mg Tablet; Drug: Glucose-Dependent Insulinotropic Polypeptide
- Placebo + GIP (Active Comparator): Placebo tablet + infusion of GIP
  Interventions: Drug: Glucose-Dependent Insulinotropic Polypeptide; Drug: Placebo Oral Tablet
- Glimepiride + GLP-1 (Active Comparator): Glimepiride + infusion of GLP-1
  Interventions: Drug: Glimepiride 1Mg Tablet; Drug: Glucagon-like Peptide-1
- Placebo + GLP-1 (Active Comparator): Placebo tablet + infusion of GLP-1
  Interventions: Drug: Glucagon-like Peptide-1; Drug: Placebo Oral Tablet
- Glimepiride + Placebo (Active Comparator): Glimepiride + infusion of placebo (saline)
  Interventions: Drug: Glimepiride 1Mg Tablet; Drug: Placebo infusion
- Placebo + Placebo (Placebo Comparator): Placebo tablet + infusion of placebo (saline)
  Interventions: Drug: Placebo Oral Tablet; Drug: Placebo infusion

INTERVENTIONS:
Drug: Glimepiride 1Mg Tablet — Glimepiride
  Arms: Glimepiride + GIP; Glimepiride + GLP-1; Glimepiride + Placebo
Drug: Glucagon-like Peptide-1 — GLP-1 infusion
  Arms: Glimepiride + GLP-1; Placebo + GLP-1
Drug: Glucose-Dependent Insulinotropic Polypeptide — GIP-infusion
  Arms: Glimepiride + GIP; Placebo + GIP
Drug: Placebo Oral Tablet — Placebo
  Arms: Placebo + GIP; Placebo + GLP-1; Placebo + Placebo
Drug: Placebo infusion — Placebo (saline)
  Arms: Glimepiride + Placebo; Placebo + Placebo

SUMMARY:
The most prevalent monogenetic diabetic subtype is named maturity onset diabetes of the young type (MODY3) or hepatocyte nuclear factor 1α (HNF1A)-diabetes. The aim of this study is to evaluate the effects of supra-physiological levels of GIP and GLP-1, respectively, on insulin and glucagon secretion at fasting plasma glucose (FPG) and "post-prandial" PG levels (1.5 × FPG) in patients with HNF1A-diabetes and matched healthy controls treated with or without a low dose of glimepiride (sulphonylurea). In addition, we will evaluate the maximal insulin and glucagon secretory capacity in both groups.

DETAILED DESCRIPTION:
A total of 6 experimental days will be performed. The following is an outline of an experimental day:

Participants will meet after a 10-hour fast. A tablet of glimepiride 1.0 mg or placebo will be administered 90 minutes before the initiation of the experiment (-90 minutes) The mean FPG will be calculated from blood samples -105, -100 and -90 minutes. Two intravenous cannulas will be inserted in a cubital vein of each arm. One intravenous cannula will be used for infusions of glucose, arginine and GIP and the other will be used to collect venous blood. The forearm from which blood samples are drawn will be placed in a heating pad (50°C) throughout the experiment for arterialisation of venous blood.

At time 0 minutes, a glucose clamp will be established at the FPG level for 60 minutes and hereafter a post-prandial clamp period of 1.5 × FPG for another 60 minutes. At time 120 minutes, a bolus of 5g of L-arginine (given as 50% arginine HCl) will be infused during 30 seconds. The post-prandial clamp will be maintained for another 10 minutes until time 130 minutes to prevent reactive hypoglycaemia. Throughout the experiment (0-130 minutes) a continuous infusion of either GIP (1.5 pmol/kg/min), GLP-1 (0.5 pmol/kg/min) or placebo (saline) will be administered.

During the experiment PG will be kept stable by a continuous 20%-glucose infusion. The rate of infusion will be regulated according to PG determined by bed-site measurements every 5 minutes. After 60 minutes, a post-prandial clamp will be established by a bolus infusion over one minute using 50%-glucose to target 1.5 × FPG (the amount of glucose to be administered will calculated as follows: (1.5 × FPG - FPG) × 35 mg glucose × weight in kilogram).

ELIGIBILITY:
Participants

Ten patients with HNF1A-diabetes and ten matched healthy controls will be recruited. Different inclusion and exclusion criteria applies for the two groups:

Inclusion criteria for HNF1A-patients

* Patients with HNF1A-diabetes verified by genetic testing
* Patients treated with diet or sulphonylurea monotherapy
* Normal haemoglobin (males 8.3-10.5 mmol/l, females 7.3-9.5 mmol/l)
* Informed consent

Exclusion criteria for HNF1A-patients

* Nephropathy (estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2 and/or albuminuria)
* Liver disease (serum alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) above 2 × normal values)
* Pregnancy or breastfeeding

Inclusion criteria for healthy controls

* FPG ≤6 mmol/l and glycated haemoglobin (HbA1c) ≤43 mmol/mol
* Normal haemoglobin as defined above
* Age ≥18 years
* Informed consent

Exclusion criteria for healthy controls

* No family history of type 1 or type 2 diabetes
* Nephropathy (defined above)
* Liver disease (defined above)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Insulin secretion | 0-120 minutes
  Incremental area under the curve (iAUC) for insulin (measured as C-peptide) at time 0-60 minutes, time 60-120 minutes and time 0-120 minutes

SECONDARY OUTCOMES:
Glucagon secretion | 0-120 minutes
  Incremental area under the curve (iAUC) for plasma glucagon at time 0-60 minutes, time 60-120 minutes and time 0-120 minutes
Maximal insulin secretion | 120-125 minutes
  Arginine maximal insulin secretion test.
Maximal glucagon secretion | 120-125 minutes
  Arginine maximal glucagon secretion test.
Amount glucose used to maintain the glucose clamp | 0-120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Christensen AS, Haedersdal S, Storgaard H, Rose K, Hansen NL, Holst JJ, Hansen T, Knop FK, Vilsboll T. GIP and GLP-1 Potentiate Sulfonylurea-Induced Insulin Secretion in Hepatocyte Nuclear Factor 1alpha Mutation Carriers. Diabetes. 2020 Sep;69(9):1989-2002. doi: 10.2337/db20-0074. Epub 2020 Jun 9. PMID 32518064